CLINICAL TRIAL: NCT07391930
Title: Efficacy of a High-Intensity Interval Training Program and Analysis of Menstrual Health Experience in Women With Primary Dysmenorrhea: A Mixed-Methods Randomized Controlled Trial.
Brief Title: High-Intensity Interval Training and Menstrual Health Experience in Primary Dysmenorrhea.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Esther María Pindado Pérez, PhD Student, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPP-2026
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Dysmenorrhea Primary; Menstrual Pain; Pelvic Pain
Keywords: High- Intensity Interval Training; Quality of Life; Menstrual Health; Therapeutic Exercise
MeSH Terms: conditions — Dysmenorrhea; Pelvic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Interval Training as Therapeutic Exercise + Menstrual Health Education Workshop (Experimental): Participants in this arm will receive a 2-hour online menstrual health education workshop and will perform 2 sessions per week of supervised online High-Intensity Interval Training (HIIT) for 12 weeks. They will also complete weekly qualitative diaries.
  Interventions: Behavioral: Supervised Online HIIT Program; Behavioral: Menstrual Health Workshop
- Menstrual Health Education Workshop (Active Comparator): Participants in this arm will receive the same 2-hour online menstrual health education workshop and will complete the same weekly qualitative diaries, but will not perform the HIIT program during the 12-week study period.
  Interventions: Behavioral: Menstrual Health Workshop

INTERVENTIONS:
Behavioral: Supervised Online HIIT Program — The intervention consists of a total of 24 exercise sessions delivered over 12 weeks (frequency: 2 sessions per week). Each session is conducted online and supervised in real-time by a physical therapist. The 24 sessions follow a structured progression of high-intensity intervals, separated by active recovery periods.
  Arms: High-Intensity Interval Training as Therapeutic Exercise + Menstrual Health Education Workshop
Behavioral: Menstrual Health Workshop — A 2-hour online educational session covering menstrual cycle physiology, pain neurophysiology, and self-care strategies. This intervention aims to improve menstrual health literacy and provide tools for pain self-management

SUMMARY:
The goal of this study is to evaluate whether a 12-week online supervised high-intensity interval training program can reduce menstrual pain and improve quality of life in women with primary dysmenorrhea. Participants will be divided into two groups: one receiving an educational workshop and the HIIT program, and a control group receiving only the workshop. Additionally, the study seeks to understand the personal experience of these women through weekly health diaries, exploring how the intervention affects their relationship with their bodies and their menstruation. The ultimate goal is to offer new, non-pharmacological evidence-based tools for managing menstrual pain.

DETAILED DESCRIPTION:
This research follows a convergent mixed-methods design integrating a randomized controlled trial with a descriptive qualitative study.

Fifty women (aged 18-40) with primary dysmenorrhea will be randomized into two arms:

Experimental Group: 12 weeks of online supervised HIIT (2 sessions/week) plus a menstrual health educational workshop.

Control Group: Menstrual health educational workshop only. Clinical variables (pain intensity via NRS, quality of life via SF-12, and pain characteristics via McGill Questionnaire) will be collected at baseline, 3 months (post-intervention), and 6 months (follow-up).

Simultaneously, all participants will complete a weekly semi-structured digital diary for 12 weeks. These diaries are designed to capture the "thick description" of their menstrual health experience, focusing on the evolution of their relationship with their body and menstruation, perceptions of self-management and empowerment and barriers and facilitators for adherence to the exercise program (in the experimental group).

Following the convergent design, quantitative statistical results will be integrated with the thematic analysis of the diaries. This merging of data will provide a holistic understanding of how high-intensity exercise influences not only physical symptoms but also the biopsychosocial perception of menstrual health in young women.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous
* primary dysmenorrhea
* body mass index between 18 and 30
* menstrual pain >5 according to the Numeric Pain Scale
* exercise >45 minutes/week
* understand Spanish and can freely read and sign the informed consent form

Exclusion Criteria:

* amenorrhea or cycles >35 days
* secondary dysmenorrhea
* pelvic or abdominal surgical intervention
* use of hormonal drugs
* diagnosed with fibromyalgia, muscoloskeletal injuries or medical comorbidities that prevent them from performing intense exercise
* receiving physiotherapy for pelvic floor disorders
* intense exercise >75 minutes/week

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Change in Menstrual Pain Intensity | Baseline (Month 0), Post-intervention (Month 3), and Follow-up (Month 6, Month 9)
  Measured using the Numeric Rating Scale (NRS), where 0 represents "no pain" and 10 represents "the worst pain imaginable." Participants will report their peak pain intensity during their menstrual period.

SECONDARY OUTCOMES:
Health-Related Quality of Life | Baseline (Month 0), Post-intervention (Month 3), and Follow-up (Month 6, Month 9)
  Assessed using the Short Form-12 (SF-12) Health Survey, which measures physical and mental health components. Higher scores indicate better quality of life.
Participant Menstrual Health Experience and Self-Management. | Weekly during the 12-week intervention period
  Qualitative assessment through the thematic analysis of weekly semi-structured digital diaries. This measure explores the evolution of the participants' relationship with their bodies, the practical application of self-care strategies, and the subjective perception of the intervention's impact. Data will be analyzed using a phenomenological approach to identify emerging themes.
Quality of Sleep | Baseline (Month 0), Post-intervention (Month 3), and Follow-up (Month 6, Month 9)
  Assessed using the Pittsburgh Sleep Quality Index (PSQI). It measures seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Scores range from 0 to 21, where higher scores indicate poorer sleep quality.
Levels of Depression, Anxiety, and Stress | Baseline (Month 0), Post-intervention (Month 3), and Follow-up (Month 6, Month 9).
  Measured using the Depression, Anxiety, and Stress Scale (DASS-21). This 21-item scale provides independent scores for each of the three psychological states. Higher scores reflect higher levels of distress.
Work Productivity and Activity Impairment | Baseline (Month 0), Post-intervention (Month 3), and Follow-up (Month 6, Month 9).
  Measured using the Work Productivity and Activity Impairment (WPAI) questionnaire. It evaluates the impact of menstrual pain on work absenteeism, presenteeism, and daily activity impairment. Results are expressed as percentages of impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Navarro Brazalez, PhD, Study Director — Universidad de Alcala
Locations (1):
- Universidad de Alcalá, Facultad de Enfermeria y Fisioterapia, Alcalá de Henares, Madrid, Spain